CLINICAL TRIAL: NCT03800108
Title: Stimulation Parameters and Non-motor Symptoms in PD Treated With DBS
Acronym: FREQUENCY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped early due to insufficient staff to continue EEG data collection and analysis following the departure of key study personnel.
Sponsor: Darlene Floden (Other)
Responsible Party: Sponsor-Investigator, Darlene Floden, Staff Neuropsychologist, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-1350
Record Dates: First submitted 2018-05-23; First posted 2019-01-11 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized DBS adjustments (Other): Individualized stimulation adjustments based on pre- and post- DBS implantation MRIs
  Interventions: Procedure: Personalized DBS adjustments

INTERVENTIONS:
Procedure: Personalized DBS adjustments — Individualized stimulation adjustments based on pre- and post- DBS implantation MRIs

SUMMARY:
This study evaluates the role of subthalamic nucleus (STN) stimulation location and frequency on a range of cognitive processes in Parkinson's patients who have undergone Deep Brain Stimulation (DBS).

DETAILED DESCRIPTION:
Pre- and post- DBS implantation brain scans will be reviewed by the study team to see if patients' DBS settings can be personalized. If so, study subjects will undergo adjustments to their DBS settings and be asked to perform cognitive tests. Some patients will be asked to come back for a second visit for brain scans.

ELIGIBILITY:
Inclusion Criteria:

1. Between 40 and 70 years of age,
2. Ability to provide informed consent,
3. Clinical diagnosis of idiopathic Parkinson disease (PD) by a movement disorders neurologist,
4. Disease duration of at least 4 years,
5. Treated with bilateral STN DBS for at least 3 months prior to study enrollment.

Exclusion Criteria:

1. History of prior neurosurgical intervention for PD (e.g., DBS, thalamotomy, pallidotomy)
2. History of other central nervous system disease (excluding migraine),
3. Presence of active psychiatric symptoms meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for Axis-I disorder on formal psychiatric evaluation, with the exception of mild depression (Beck Depression Inventory-2 score below 19),
4. Cognitive impairment meeting Diagnostic and Statistical Manual of Mental Disorders-4th Edition (DSM-IV) criteria for dementia on formal neuropsychological evaluation,
5. Current alcohol or substance abuse,
6. Lack of fluency in English which would invalidate cognitive testing,
7. Hearing or visual impairment precluding cognitive testing.

   Exclusion criteria for Day 2 procedures:
8. Inability to safely undergo MRI procedure (i.e., metal objects like prostheses, pacemakers)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darlene Floden, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five participants were enrolled from 05/30/2018 to 11/04/2019.
Pre-assignment Details: Following enrollment, participants completed a washout period by withholding Parkinson's medications overnight before each study session to reduce confounding effects. EEG electrodes were then applied prior to cognitive and motor testing under varied deep brain stimulation (DBS) parameters. No participants were excluded after enrollment. Key personnel changes led to early study closure, limiting the final data collection.
Period: Overall Study
Arm/Group | Personalized DBS Adjustments
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Personalized DBS Adjustments
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time
Description: Subjects will complete one or more measures of cognitive processing requiring speeded responses to stimuli. Changes in reaction time will be compared to 'off stimulation'
Time Frame: 30-60 minutes after stimulation adjustment
Measure: Count of Participants; unit: Participants
Arm/Group | Personalized DBS Adjustments
Number analyzed (Participants) | 3
Participants
  Inhibitory control worse with Ventral High Hz | 2
  Inhibitory control worse with Dorsal Low Hz | 1

2. Primary Outcome: Verbal Fluency
Description: Change in the number words that patients generate to letter or semantic category cues will be compared to 'off stimulation'
Time Frame: 30-60 minutes after stimulation adjustment
Population: Patients with Deep Brain Stimulation Electrodes implanted to treat Parkinson's disease
Measure: Mean (Full Range); unit: words
Arm/Group | Personalized DBS Adjustments
Number analyzed (Participants) | 3
words
  Change at Dorsal High Hz | 6.3 [2 to 11]
  Change at Ventral Low Hz | -0.3 [-5 to 5]

3. Primary Outcome: Finger Tapping Speed
Description: Change in upper extremity speed (# of taps in 10 seconds) will be compared to 'off stimulation'
Time Frame: 30-60 minutes after stimulation adjustment
Measure: Mean (Full Range); unit: finger taps
Arm/Group | Personalized DBS Adjustments
Number analyzed (Participants) | 3
finger taps
  Taps change at Dorsal High Hz | 2.1 [-1 to 5]
  Taps change at Ventral Low Hz | 2.2 [.66 to 4.5]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 2-3 days, depending on the number of study sessions, with monitoring by Clinical Research Unit (CRU) nursing staff and the research team. Participants were assessed for safety and well-being after each change in stimulation parameters during EEG recording and fMRI sessions as well as by telephone one day after their final study session.
Arm/Group | Personalized DBS Adjustments
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
Limitations of this trial include early termination due to a lack of eligible patients which led to a reduced sample size and limited data collection. This constraint impacted the statistical power and the ability to conduct complete analyses as initially planned. Additionally, technical limitations related to EEG data collection and analysis emerged, as key personnel responsible for EEG recording and data processing were unavailable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03800108/Prot_SAP_000.pdf